CLINICAL TRIAL: NCT06601985
Title: Exploring the Effect of Applying Colonic J-pouch Forming in Anorectal Preservation Surgery for Ultra-low Rectal Cancer on Postoperative Bowel Control Function
Brief Title: Exploring the Effect of Colonic J-pouch in Anorectal Preservation Surgery for Ultra-low Rectal Cancer.
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Feng-Min, Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: 24K30
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectum Cancer; Faecal Incontinence; Faecal Incontinence with Faecal Urgency; Low Anterior Resection Syndrome; Leakage, Anastomotic
MeSH Terms: conditions — Rectal Neoplasms; Encopresis; Low Anterior Resection Syndrome; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- J-pouch anastomosis group: Patient with ultra-low rectal cancer undergoing Sphincter- preserving surgery with one-stage anastomosis using a colon J-pouch.
  Interventions: Procedure: J-pouch anastomosis
- direct anastomosis group: Patient with ultra-low rectal cancer undergoing Sphincter- preserving surgery with one-stage direct anastomosis.
  Interventions: Procedure: direct anastomosis

INTERVENTIONS:
Procedure: J-pouch anastomosis — Patient with ultra-low rectal cancer undergoing Sphincter- preserving surgery with one-stage anastomosis using a colon J-pouch.
  Groups: J-pouch anastomosis group
Procedure: direct anastomosis — Patient with ultra-low rectal cancer undergoing Sphincter- preserving surgery with one-stage direct anastomosis.
  Groups: direct anastomosis group

SUMMARY:
The occurrence of colorectal cancer has increased from the third most common cancer in 2018 to the second most common cancer in 2023. The practice of anal preservation surgery for ultra-low rectal cancer is being adopted gradually. Ultra-low rectal cancer patients who have undergone anal preservation are at an increased risk of developing significant bowel complications. The objective of this study was to examine the relationship between the type of bowel reconstruction following anal preservation surgery, and the subsequent outcomes of bowel function, quality of life and complication rates in patients with ultra-low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of intestinal cancer, with the lower edge of the tumour <5 cm from the anus or <3 cm from the dentate line, and treated with anus-preserving surgery;
2. No distant metastasis;
3. Age >18 years old;
4. Voluntary enrollment in the study and signing of an informed consent.

Exclusion Criteria:

1. A combination of severe cardiopulmonary, hepatic, renal, and other underlying diseases with a greater anaesthetic risk (ASA ≥ grade 4);
2. preoperative anal stenosis and anal nonfunction;
3. temporary stoma diversion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population is the patients who diagnosed as ultra-low rectal adenocarcinoma cases by preoperative pathology and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-03-11 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
LARS score | From 1 month postoperatively to 12 months postoperatively
  The LARS scale has five questions with a total score of 42. A score of 0-20 lacks diagnostic value for LARS, while a score of 21-29 indicates mild LARS and a score above 29 indicates major LARS.
FIQL | From 1 month postoperatively to 12 months postoperatively
  The FIQL is a specific quality-of-life assessment scale applicable to the symptoms of colorectal cancer patients. It comprises 29 items, which are divided into four dimensions: lifestyle (10 items), coping/behavior restriction(9 items), depression/self-perception (7 items), and embarrassment (3 items).
Vaizey score | From 1 month postoperatively to 12 months postoperatively
  The Wexner scale has five parts with a total score of 20, while the Vaizey scale is further refined on the basis of Wexner and has seven parts with a total score of 24. Higher scores on these scales indicate poorer anal functioning.
Wexner score | From 1 month postoperatively to 12 months postoperatively
  The Wexner scale has five parts with a total score of 20, while the Vaizey scale is further refined on the basis of Wexner and has seven parts with a total score of 24. Higher scores on these scales indicate poorer anal functioning.

SECONDARY OUTCOMES:
Surgical complications | From 1 month postoperatively to 12 months postoperatively
  Records post-operative anastomotic fistula, infection, bleeding, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Le Zhuang, MD, PhD, Study Chair — Shanghai Tenth People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Yanchang Road, Jing'an District, Shanghai, China, Shanghai, Jingan, China

IPD SHARING:
Plan to Share IPD: Undecided